CLINICAL TRIAL: NCT01603589
Title: Research on Remote End-organ Protection, Clinical Outcome and Quality of Life With Implementation of the Novel Minimal Extracorporeal Circulation Circuit in Open Heart Surgery
Brief Title: Comparison of Minimal Versus Conventional Extracorporeal Circulation in Coronary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHEPA_CTS_04
Record Dates: First submitted 2012-05-21; First posted 2012-05-22 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Bypass
Keywords: coronary artery disease; coronary artery bypass grafting; cardiopulmonary bypass; minimal extracorporeal circulation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MiECC group (Active Comparator): Patients operated for elective coronary artery bypass grafting with the use of minimal invasive extracorporeal circulation (MiECC).
  Interventions: Procedure: Coronary artery bypass grafting with the use of minimal invasive extracorporeal circulation
- CECC group (Active Comparator): Patients operated for elective coronary artery bypass grafting under conventional extracorporeal circulation (CECC).
  Interventions: Procedure: Coronary artery bypass grafting under conventional extracorporeal circulation

INTERVENTIONS:
Procedure: Coronary artery bypass grafting with the use of minimal invasive extracorporeal circulation — We use a prototype AHEPA (modular type IV) circuit comprised of the standard and a standby accessory. Components of the standard circuit include: aortic cannula, three-stage venous cannula, coated tubing, a centrifugal pump, a new-generation membrane oxygenator with integrated arterial filter, a venous air removal device, a soft coated bag and pulmonary artery as well as aortic root vent. In addition, there is a standby hard-shell reservoir in parallel to the venous line, so as to convert the closed system to an open one. The standby component is bridged to the main circuit with an afferent line which is connected just before the VARD sending blood to the hard-shell reservoir and an efferent that re-directs it back to the VARD. A cell-saver device is added to the circuit for collecting shed blood and washing red blood cells for autotransfusion.
  Arms: MiECC group
Procedure: Coronary artery bypass grafting under conventional extracorporeal circulation — A standard open CPB circuit is used, consisting of uncoated PVC tubing, a hard-shell venous reservoir, a microporous membrane oxygenator (Dideco, Mirandola, Italy) and a roller pump (Stöckert S3, Munich, Germany). The circuit contains a 40 μm arterial line blood filter (Dideco, Mirandola, Italy) and it is primed with 1500 mL of a balanced crystalloid/colloid solution (1000 mL of Ringer's solution, 200 mL of mannitol 20%, and 300 mL of hydroxyethyl starch 6%). Cardiotomy as well as sump sucker are integrated to the circuit.
  Arms: CECC group

SUMMARY:
The aim of this study is to assess the effect of minimal (MiECC) versus conventional (CECC) extracorporeal circulation on perfusion characteristics and remote end-organ protection (lungs, brain, kidneys, liver, stomach, intestine), after elective coronary bypass grafting (CABG).

DETAILED DESCRIPTION:
The aim of this study is to investigate whether coronary surgery with minimal Invasive Extracorporeal Circulation (MiECC) offers advantage over conventional CPB (CECC). In order to draw an evidence-based conclusion, the investigators aim to evaluate perfusion characteristics during coronary surgery with MECC and associated remote end-organ function. Improved end-organ protection translates into improved clinical outcome which greatly affects quality of life. This is the first study in the literature adequately powered to analyse organ pathophysiology during surgery with MECC and at the same time correlating common clinical variables with a detailed quality of life evaluation. Superiority of MECC could provide firm evidence towards widespread use of MECC in coronary surgery as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective coronary artery bypass grafting

Exclusion Criteria:

* history of psychiatric disorder
* inability to undergo neuropsychological assessment
* history of transient ischemic attack or stroke
* carotid artery stenosis > 60% assessed by duplex ultrasonography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Remote end-organ perfusion and function (brain, lungs, liver, kidneys, stomach, intestine) intraoperatively and postoperatively during hospital stay | 30 days
  Remote end-organ perfusion and function at 30 days follow-up after elective coronary artery bypass grafting with the use of minimal (MiECC) versus conventional (CECC) extracorporeal circulation.

SECONDARY OUTCOMES:
Postoperative major adverse cardiac and cerebrovascular events (MACCE) that comprise: myocardial infarction, low cardiac output syndrome, stroke, renal failure. | 30 days
  Postoperative major adverse cardiac and cerebrovascular events (MACCE) that comprise: myocardial infarction, low cardiac output syndrome, stroke, renal failure at 30 days follow-up after elective coronary artery bypass grafting with the use of minimal (MiECC) versus conventional (CECC) extracorporeal circulation.
Duration of mechanical ventilation | 30 days
  Duration of mechanical ventilation at 30 days follow-up after elective coronary artery bypass grafting with the use of minimal (MiECC) versus conventional (CECC) extracorporeal circulation.
Length of ICU stay | 30 days
  Length of ICU stay at 30 days follow-up after elective coronary artery bypass grafting with the use of minimal (MiECC) versus conventional (CECC) extracorporeal circulation.
Development of new postoperative atrial fibrillation. | 30 days
  Development of new postoperative atrial fibrillation at 30 days follow-up after elective coronary artery bypass grafting with the use of minimal (MiECC) versus conventional (CECC) extracorporeal circulation.
Neurocognitive function | 6 months postoperatively
  Neurocognitive evaluation with a battery of specialized tests performed by a dedicated and experienced team in clinical psychology. Evaluation will be performed at specific time intervals: preoperatively, at 1-, 3- and 6-month follow-up.
Health-related quality of life | 6 months postoperatively
  Change in quality of life assessed with SF-36 questionnaire after coronary artery bypass grafting with minimal versus conventional extracorporeal circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, PhD, FETCS, Principal Investigator — Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece
Locations (1):
- Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Anastasiadis K, Antonitsis P, Haidich AB, Argiriadou H, Deliopoulos A, Papakonstantinou C. Use of minimal extracorporeal circulation improves outcome after heart surgery; a systematic review and meta-analysis of randomized controlled trials. Int J Cardiol. 2013 Apr 5;164(2):158-69. doi: 10.1016/j.ijcard.2012.01.020. Epub 2012 Feb 8. PMID 22325958
- [Background] Anastasiadis K, Asteriou C, Deliopoulos A, Argiriadou H, Karapanagiotidis G, Antonitsis P, Grosomanidis V, Misias G, Papakonstantinou C. Haematological effects of minimized compared to conventional extracorporeal circulation after coronary revascularization procedures. Perfusion. 2010 Jul;25(4):197-203. doi: 10.1177/0267659110373840. Epub 2010 Jun 1. PMID 20515982
- See also: CardioThoracic Surgery Network — http://www.ctsnet.org